CLINICAL TRIAL: NCT07265791
Title: Multicenter, Randomized, Subject & Independent Evaluator-blind, Matched Pairs, Active-controlled, Non-inferiority, Pivotal Study to Evaluate the Efficacy and Safety of Injection With JTM104 as Compared to Juvederm® ULTRA PLUS XC in Temporary Correction of Moderate to Severe Nasolabial Folds
Brief Title: Study of JTM104 Injection vs. Juvederm in Treating Moderate to Severe Nasolabial Folds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jetema Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JT-D-104-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Nasolabial Folds, Wrinkles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTM104 (Experimental): HA Filler
  Interventions: Biological: JTM104
- Juvederm® ULTRA PLUS XC (Active Comparator): HA Filler
  Interventions: Biological: Juvederm® ULTRA PLUS XC

INTERVENTIONS:
Biological: JTM104 — JTM104 contains 22.8 mg/mL cross-linked hyaluronic acid, 1.2 mg/mL hyaluronic acid, and 3 mg/mL lidocaine. The product will be injected into the nasolabial folds, with a maximum volume of 1 mL per side.
  Arms: JTM104
Biological: Juvederm® ULTRA PLUS XC — Juvederm® ULTRA PLUS XC contains 22.8 mg/mL cross-linked hyaluronic acid, 1.2 mg/mL hyaluronic acid, and 3 mg/mL lidocaine. The product will be injected into the nasolabial folds, with a maximum volume of 1 mL per side.
  Arms: Juvederm® ULTRA PLUS XC

SUMMARY:
Study of JTM104 Injection vs. Juvederm in Treating Moderate to Severe Nasolabial Folds

DETAILED DESCRIPTION:
Multicenter, Randomized, Subject & Independent Evaluator-blind, Matched pairs, Active-controlled, Non-inferiority, Pivotal study to evaluate the Efficacy and Safety of Injection with JTM104 as Compared to Juvederm® ULTRA PLUS XC in temporary correction of Moderate to Severe Nasolabial folds

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 75 years
* Voluntarily provided written informed consent
* Moderate to severe symmetrical nasolabial folds (WSRS score 3 or 4 on both sides)
* Agree to discontinue other facial dermatologic treatments (e.g., fillers, botulinum toxin, laser) during the study
* Able to understand instructions and comply with study procedures

Exclusion Criteria:

* Untreated scars or facial skin infections/diseases affecting the mid/lower face within the past year
* History of severe allergy or hypersensitivity to device components
* Facial invasive procedures within the past 6 months (including surgery, laser, botulinum toxin)
* Use of certain medications (anticoagulants, immunosuppressants, steroids) within specified washout periods
* Participation in other interventional clinical trials within 4 weeks before screening or during study
* Non-compliance with contraception requirements or pregnancy/lactation during study
* Deemed unsuitable by investigator for any other reason

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
AE | From adverse event onset through resolution or stabilization, up to 30 days post-study completion
  Continuous follow-up of adverse events until resolution, stabilization, or cause identification; includes 30-day follow-up after study completion if unresolved.
SAE | From adverse event onset through resolution or stabilization, up to 30 days post-study completion
  Continuous follow-up of adverse events until resolution, stabilization, or cause identification; includes 30-day follow-up after study completion if unresolved.
Solicited local AE | Within 2 weeks after device application
  Local adverse events occurring at the application site within 2 weeks after device use, including pain, swelling, redness, bruising, and other injection site reactions.

OTHER OUTCOMES:
Lidocaine-Related AE | Within 30 minutes after device application
  Adverse events related to lidocaine occurring within 30 minutes after device application, including hypersensitivity, shock, and toxicity symptoms.

IPD SHARING:
Plan to Share IPD: No